CLINICAL TRIAL: NCT03661372
Title: Telesimulation and Behavioral Health: Assessment of the Integration of the Abbreviated Checklist Contextual Interview Observation Form-Adult (CIOF-A) as a Learning Tool in Interprofessional Practice & Education: A Pilot Study
Brief Title: Telesimulation and Behavioral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Northwest University of Health Sciences (Other)
Collaborators: American Association of Colleges of Osteopathic Medicine - AACOM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-020
Record Dates: First submitted 2018-08-24; First posted 2018-09-07 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Self Efficacy

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-Face (Active Comparator): Face-to-Face Group: At the beginning of the session self-efficacy will be measured. This group will receive an instructor-led 45 minute long lecture on how to evaluate work, love, and play behavioral health form on a standardized patient. A face-to- face standardized patient scenario will test the participant on the application of work, love, and play assessment. In this scenario, the participant will meet a standardized patient in the exam room to discuss a behavioral health concern. At the end of each session (approximately 2 hours later), self-efficacy will be measured.
  Interventions: Other: Face-to-face
- Robot (Active Comparator): Robot Group: At the beginning of the session self-efficacy will be measured. This group will receive an instructor-led 45 minute long lecture on how to evaluate work, love, and play behavioral health form on a standardized patient. A robot (telesimulated) standardized patient scenario will test the participant on the application of work, love, and play assessment. In this scenario, the participant will meet a standardized patient in the exam room via a robot to discuss a behavioral health concern. At the end of each session (approximately 2 hours later), self-efficacy will be measured.
  Interventions: Other: Robot

INTERVENTIONS:
Other: Robot — Use of a telesimulation robot using contextual interview format.
  Arms: Robot
Other: Face-to-face — Use of face-to-face patient interview using contextual interview format.
  Arms: Face-to-Face

SUMMARY:
This study proposes to assess attitudes, perceived proficiency, and knowledge related to telemedicine by implementing telesimulation behavioral health scenarios in a cohort of healthcare students using the Contextual Interview Observation Form.

DETAILED DESCRIPTION:
According to Mental Health America, 1 in 5 adults have a mental health condition. Mental health is associated with higher incidence of chronic diseases, lower use of medical care, and one of five most costly conditions in the US in 2006 according to the American Psychological Association. The Accreditation Council for Graduate Medical Education (ACGME) has called for residents to develop an understanding of social-behavioral sciences as a basis for patient care. ACGME advises that the curriculum is extended to physical aspects of patient care as well as the emotional, social and behavioral aspects. The Society of Teachers of Family Medicine (STFM) has also suggested the importance of the psychosocial realm. According to both the ACGME and STFM, being able to glean the necessary information is an integral part of being a family doctor.

The need for healthcare providers, medical students, and residents to possess basic interviewing, counseling and agenda setting skills to ascertain the pertinent contextual (e.g., familial, social, cultural, spiritual, etc.), health behavior, and health risk factors of patients' lives, is vital to close the gap on behavioral health and chronic diseases. In order to evaluate learners' interviewing skills, the Contextual Interview Observation Form (CIOF) an observation tool was developed using Robinson, Gould, and Strosahl's (2010) interview format. The CIOF can be used to teach a contextual interview "procedure" that is organized in a logical manner with a practical format. This "contextual interview" provides a no-cost format for the learner to capture the context of patients' behaviorally influenced health concerns and is applicable during the 4-year curriculum as well as during the clerkship years.

Many Americans lack access to health care, with an even greater shortage of access to mental health providers, especially in rural and underserved areas. Improving access to behavioral health providers and recognition of mental illness via telemedicine, could lead to improved patient outcomes and cost. However, in the pedagogical course of medical education, the investigators do not provide a robust platform for teaching telemedicine. Implementing the CIOF in a telesimulation format will allow for healthcare providers, behavior health providers, medical students, and residents to practice and experience providing basic interviewing and counseling via telemedicine. According to McCoy et al, telesimulation is "a process by which telecommunication and simulation resources are utilized to provide education, training, and/or assessment to learners at an off-site location. Off-site location refers to a distant site that would preclude the education, training, and/or assessment without the use of telecommunication resources."

Pacific Northwest University of Health Sciences educates and trains healthcare professionals emphasizing service among rural and medically underserved communities throughout the Northwest. Specifically, the investigators cover rural and underserved areas in Alaska, Washington, Oregon, Montana, and Idaho. PNWU's envisioned Institute for Interprofessional Practice & Education (IIPE) focuses on cultivating healthcare teams from a variety of professional backgrounds to enhance person-centered health care. One goal of PNWU's strategic plan is to expand graduate level educational opportunities. In response to that goal, the Yakima Valley Interprofessional Practice and Education Collaborative (YVIPEC) was established in the fall of 2014 to promote the highest quality health care in the region through a culture of inclusive and collaborative interprofessional education, practice, and scholarship. Interprofessional education (IPE) fosters a team-based approach to health care which is the approach used in rural health clinics and is reported to be critical to success in working in medically underserved areas. These collaborations include:

* Pacific Northwest University of Health Sciences (PNWU), Doctor of Osteopathic Medicine;
* Heritage University (HU), Physician Assistant Program and Nursing Program;
* Washington State University (WSU), Nursing Program and Pharmacy Program;
* Central Washington University (CWU), Paramedicine Program and Dietetics Program;
* Washington State Allied Health Center of Excellence, located at Yakima Valley College

The current PNWU College of Osteopathic Medicine (COM) curriculum includes CLIN 618, which is a second year requirement and presents a multidimensional approach to the understanding of the most common clinical entities in psychiatry and behavioral medicine. Third and fourth year courses includes BEHCS 701 Behavioral Medicine rotation which is designed for students to learn and practice skills necessary for working with patients in a mental health setting. Incorporating the COIF via telesimulation would give students, residents, and faculty the experience for use beyond course requirements and prepare them for the future of healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Any enrolled student at a participating program in the Yakima Valley Interprofessional Collaborative
* Age 18-33 (focusing on the Millennial Generation)

Exclusion Criteria:

* Able to read, write, and speak English due to the pilot nature of the study
* Have no pending litigation with any education entity within the YVIPEC

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Changes in Self-Efficacy in Patient Centeredness Questionnaire (SEPCQ27) 27-item | Baseline and approximately 2-hours after baseline
  The SEPCQ is designed to measure confidence levels at delivering patient-centered care (A 7-point Likert scale was used with "0" (to a very low degree) and "6" (To a very high degree)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Munoz, MPH, Principal Investigator — Pacific Northwest University of Health Sciences
Locations (1):
- Pacific Northwest University of Health Sciences, Yakima, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Accreditation Council for Graduate Medical Education (ACGME). (2014, July 1). ACGME program requirements for graduate medical education in family medicine. Retrieved from http://www.acgme.org/acgmeweb/Portals/0/PFAssets/Program Requirements/120_family_medicine_07012014.pdf
- [Background] Schirmer, J. M., Taylor, D., & Zylstra, R. (2008). New Set of Core Principles of Behavioral Medicine. Society of Teachers of Family Medicine.
- [Background] Robinson, P. J., Gould, D. A., & Strosahl, K. D. (2010). Real behavior change in primary care: Improving patient outcomes & increasing job satisfaction. Oakland, CA: New Harbinger Publications, Inc.
- [Background] McCoy CE, Sayegh J, Alrabah R, Yarris LM. Telesimulation: An Innovative Tool for Health Professions Education. AEM Educ Train. 2017 Feb 17;1(2):132-136. doi: 10.1002/aet2.10015. eCollection 2017 Apr. PMID 30051023
- [Background] Miller, W. R., & Rollnick, S. (2002). Motivational interviewing: Preparing people for change (2nd ed.). New York, NY: The Guilford Press.
- [Background] Berkman ND, Sheridan SL, Donahue KE, Halpern DJ, Crotty K. Low health literacy and health outcomes: an updated systematic review. Ann Intern Med. 2011 Jul 19;155(2):97-107. doi: 10.7326/0003-4819-155-2-201107190-00005. PMID 21768583
- [Derived] Rosasco J, Hanson Z, Kramer J, Steele L, Beachy B, Gothard MD, Ahmed R, McCarroll ML. A Randomized Study Using Telepresence Robots for Behavioral Health in Interprofessional Practice and Education. Telemed J E Health. 2021 Jul;27(7):755-762. doi: 10.1089/tmj.2020.0245. Epub 2020 Oct 21. PMID 33090088